CLINICAL TRIAL: NCT04720105
Title: Investigator-Initiated, Open Label Trial of a Combination of Halobetasol Propionate 0.01% Andtazarotene 0.045% Lotion (Duobrii®) for Plaque Type Psoriasis of the Hands and/or Feet
Brief Title: Combination of Halobetasol Propionate and Tazarotene Lotion (Duobrii®) for Palmoplantar Plaque Type Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Principal Investigator, Alice B Gottlieb, Clinical Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 20-0608
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Results first posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Palmoplantar Psoriasis; Plaque Psoriasis
Keywords: Palmoplantar; Psoriasis; Plaque
MeSH Terms: conditions — Psoriasis; Plaque, Amyloid | interventions — halobetasol; tazarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with plaque type psoriasis (Experimental): Participants with plaque type psoriasis to be treated with Duobrii® (halobetasol propionate 0.01%/tazarotene 0.045% lotion) to be applied thinly once a day on the affected areas of hands and/or feet.
  Interventions: Drug: Duobrii®

INTERVENTIONS:
Drug: Duobrii® — Duobrii® (halobetasol propionate 0.01%/tazarotene 0.045% lotion, HP/TAZ) will be provided at weeks 0,2,8,16 for a total of 24 weeks.
  Other Names: Halobetasol propionate 0.01%/tazarotene 0.045% lotion; HP/TAZ

SUMMARY:
The purpose of this research study is to examine the effect of Duobrii® (halobetasol propionate 0.01%/tazarotene 0.045% lotion, HP/TAZ) on plaque type psoriasis of the hands and/or feet.

DETAILED DESCRIPTION:
Plaque type psoriasis of the hands and/or feet affects approximately 3-4% of patients with psoriasis. It is characterized by well-defined erythematous desquamative plaques located on the palms and soles, which may be limited to acral involvement or occur in combination with generalized psoriasis. Psoriasis that affects the hands and/or feet has a profound impact on quality of life (QoL) as it contributes to more physical disability and discomfort than patients with other forms of psoriasis, such as difficulty walking or using the hands.

Furthermore, psoriasis of the hands and/or feet is generally considered a therapeutic challenge because the thicker stratum corneum reduces the penetration of topical treatment agents. Systemic treatments (retinoids, psoralen-ultraviolet A [PUVA], methotrexate, cyclosporine, and biologic therapy) have shown limited efficacy on psoriasis in acral areas. Unfortunately, patients with hand and/or foot involvement often have too low of body surface area (BSA) to participate in clinical trials for new psoriasis treatments, resulting in limited studies among this sub-population and no clear treatment algorithm.

The high unmet need for an effective treatment for psoriasis of the hands and/or feet has been addressed in recent years with the development of new medications for generalized psoriasis that may also be effective in treating disease localized to acral areas. In 2015, two multicenter, double-blind, randomized, parallel-group phase 3 studies were conducted to assess the safety, tolerability, and efficacy of lotion containing a combination of halobetasol propionate 0.01% and tazarotene 0.045% (HP/TAZ). The study population was subjects with moderate-to-severe psoriasis. The study results found that treatment success (defined as at least a 2-grade improvement from baseline Investigator Global Assessment score and a score of clear or almost clear) was achieved in around 40% of subjects by week 8, with substantial reductions in affected BSA, improvement in QoL, and a significant reduction in signs and symptoms of psoriasis.

These phase 3 studies did not include a sub-analysis of the effect of HP/TAZ on psoriasis of the hands and/or feet. Given that topical steroids and topical retinoids are separately recommended as treatment options for psoriasis of the hands and/or feet, an agent that safely combines these medications - and that has demonstrated safety and efficacy in generalized psoriasis - offers a potential treatment for psoriasis of the hands and/or feet.

The purpose of the study described in this protocol is to evaluate the effect of HP/TAZ on plaque type psoriasis of the hands and/or feet after 24 weeks of daily treatment. In addition, given the impact of this variant of psoriasis on QoL and the relative lack of currently available treatment options, this study will also evaluate the impact of HP/TAZ treatment on patient-reported QoL measures and treatment satisfaction scoring.

ELIGIBILITY:
Inclusion Criteria

* Subject is able to provide written, informed consent and comply with the study protocol.
* Subject is at least 18 years of age.
* Subject has a diagnosis of plaque-type palmar and/or plantar psoriasis.
* Patient has at least one psoriatic plaque outside of the palms and soles or psoriatic nail findings.
* Subject has a ppPGA ≥ 3 at screening/baseline visit.
* Subject is using adequate birth control during the study period as defined as follows:

  1. Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy; OR
  2. Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]; PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

     OR
  3. Option 3: Abstinence from sex when it is a lifestyle choice, and not just a social circumstance.

Exclusion Criteria

* Subject is not able to provide written, informed consent and comply with the study protocol.
* Subject is less than 18 years of age.
* Subject has non-plaque type psoriasis on the hands and/or feet.
* Patient does not have any evidence of psoriasis elsewhere.
* Subject has concurrent cutaneous disease affecting the hands and/or feet that would interfere with assessments.
* Subject has a ppPGA < 3 at screening/baseline visit.
* Subject refuses to discontinue concomitant prescription medications on hands and/or feet.
* Subject has used topical prescription treatments or received phototherapy treatment for psoriasis within 2 weeks of screening/baseline visit.
* Subject has used intralesional kenalog within 4 weeks of screening/baseline visit.
* Subject has taken oral treatments for psoriasis within 4 weeks of screening/baseline visit.
* Subject has received any treatment with biologic medications within 5 half-lives (if known) or 16 weeks prior to screening/baseline, whichever is longer.
* Subject refuses to use adequate birth control during the duration of the study period.
* Subject is currently pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Gottlieb, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Downtown Union Square, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Engin B, Askin O, Tuzun Y. Palmoplantar psoriasis. Clin Dermatol. 2017 Jan-Feb;35(1):19-27. doi: 10.1016/j.clindermatol.2016.09.004. Epub 2016 Sep 10. PMID 27938808
- [Background] Raposo I, Torres T. Palmoplantar Psoriasis and Palmoplantar Pustulosis: Current Treatment and Future Prospects. Am J Clin Dermatol. 2016 Aug;17(4):349-58. doi: 10.1007/s40257-016-0191-7. PMID 27113059
- [Background] Gold LS, Lebwohl MG, Sugarman JL, Pariser DM, Lin T, Martin G, Pillai R, Israel R, Ramakrishna T. Safety and efficacy of a fixed combination of halobetasol and tazarotene in the treatment of moderate-to-severe plaque psoriasis: Results of 2 phase 3 randomized controlled trials. J Am Acad Dermatol. 2018 Aug;79(2):287-293. doi: 10.1016/j.jaad.2018.03.040. Epub 2018 Apr 1. PMID 29614243
- [Background] Sugarman JL, Weiss J, Tanghetti EA, Bagel J, Yamauchi PS, Stein Gold L, Lin T, Martin G, Pillai R, Israel R. Safety and Efficacy of a Fixed Combination Halobetasol and Tazarotene Lotion in the Treatment of Moderate-to-Severe Plaque Psoriasis: A Pooled Analysis of Two Phase 3 Studies. J Drugs Dermatol. 2018 Aug 1;17(8):855-861. PMID 30124724
- [Background] Gottlieb A, Sullivan J, van Doorn M, Kubanov A, You R, Parneix A, Hugot S, Milutinovic M. Secukinumab shows significant efficacy in palmoplantar psoriasis: Results from GESTURE, a randomized controlled trial. J Am Acad Dermatol. 2017 Jan;76(1):70-80. doi: 10.1016/j.jaad.2016.07.058. Epub 2016 Oct 1. PMID 27707593
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Plaque Type Psoriasis: Participants with plaque type psoriasis to be treated with Duobrii® (halobetasol propionate 0.01%/tazarotene 0.045% lotion, HP/TAZ) to be applied thinly once a day on the affected areas of hands and/or feet at weeks 0,2,8,16 for a total of 24 weeks.
Period: Overall Study
Arm/Group | Participants With Plaque Type Psoriasis
Started | 22
Completed | 17
Not Completed | 5
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Plaque Type Psoriasis
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Palmoplantar Physician Global Assessment (ppPGA)
Description: Number of participants achieving Palmoplantar Physician Global Assessment (ppPGA) of 0 (clear) or 1 (almost clear/minimal) after 24 weeks of treatment. The ppPGA is based on the Investigators Global Assessment (IGA) modified version 11, specifically applied to the hands and/or feet: 0 (clear), 1 (almost clear/minimal), 2 (mild), 3 (moderate), 4 (marked/moderate-to-severe), 5 (severe)
Time Frame: Baseline and Week 24
Population: For week 24 data, results reported for the patients who had completed study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Plaque Type Psoriasis
Number analyzed (Participants) | 22
score on a scale
  Baseline | 3.47 (0.72)
  Week 24: number analyzed (Participants) | 17
  Week 24 | 2.24 (1.03)

2. Secondary Outcome: Dermatology Quality of Life Index (DLQI)
Description: Patient-reported outcomes evaluated by Dermatology Quality of Life Index (DLQI). DLQi is a 10-item questionnaire, each question is scored from 0 to 3, giving a possible score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life). Higher score indicates poorer health outcome.
Time Frame: Baseline and Week 24
Population: For week 24 data, results reported for the patients who had completed study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Plaque Type Psoriasis
Number analyzed (Participants) | 22
score on a scale
  Baseline | 6.24 (5.83)
  Week 24: number analyzed (Participants) | 17
  Week 24 | 4.94 (5.58)

3. Secondary Outcome: Numerical Rating Scale (NRS)
Description: Treatment satisfaction evaluated by a Numerical Rating Scale (NRS). Full scale from 0 to 10, higher score indicates poorer health outcome.
Time Frame: Baseline and Week 24
Population: For week 24 data, results reported for the patients who had completed study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Participants With Plaque Type Psoriasis
Number analyzed (Participants) | 22
score on a scale
  Baseline | 1.35 (2.18)
  Week 24: number analyzed (Participants) | 17
  Week 24 | 1.29 (2.05)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Participants With Plaque Type Psoriasis
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT04720105/Prot_SAP_000.pdf